CLINICAL TRIAL: NCT00074087
Title: Phase II Clinical Trial With Caelyx Mono-Chemotherapy in Patients With Advanced Mycosis Fungoides Stage IIb, IVa and IVb With or Without Previous Chemotherapy
Brief Title: Liposomal Doxorubicin in Treating Patients With Stage IIB, Stage IVA, or Stage IVB Recurrent or Refractory Mycosis Fungoides
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-21012; 2004-001746-32 (EudraCT Number)
Record Dates: First submitted 2003-12-10; First posted 2003-12-11 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Lymphoma
Keywords: stage II mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; stage IV cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Mycosis Fungoides; Sezary Syndrome; Lymphoma, T-Cell, Cutaneous

ARMS (1):
- Caelyx (Experimental): doxorubicin HCl liposome IV over 1 hour on days 1 and 15. Treatment repeats every 28 days for up to 6 courses.
  Interventions: Drug: pegylated liposomal doxorubicin hydrochloride

INTERVENTIONS:
Drug: pegylated liposomal doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as liposomal doxorubicin, use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of liposomal doxorubicin in treating patients who have stage IIB, stage IVA, or stage IVB recurrent or refractory mycosis fungoides.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the antitumor activity of doxorubicin HCl liposome, in terms of response rate (complete response and partial response), in patients with stage IIB, IVA, or IVB recurrent or refractory mycosis fungoides.

Secondary

* Determine the time to progression and duration of response in patients treated with this drug.
* Determine the toxicity of this drug in these patients.

OUTLINE: This is an open-label, nonrandomized, multicenter study.

Patients receive doxorubicin HCl liposome IV over 1 hour on days 1 and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity or until a maximum cumulative anthracycline(s) dose of 400 mg/m^2 has been reached (including anthracyclines from prior treatment).

Patients are followed every 12 weeks until disease progression.

PROJECTED ACCRUAL: A total of 48 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed mycosis fungoides

  * Stage IIB, IVA, or IVB
* Refractory or recurrent disease after at least 2 of the following prior therapies:

  * Local and/or systemic steroids
  * Retinoids
  * Interferon alfa
  * Local carmustine
  * Systemic chemotherapy
  * Psoralen and ultraviolet A (PUVA) light therapy
* No CNS involvement
* No erythroderma (T4)

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* Neutrophil count at least 1,500/mm^3
* WBC at least 2,000/mm^3
* Platelet count at least 75,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT and SGPT no greater than 2.5 times ULN

Renal

* Creatinine no greater than 1.5 times ULN

Cardiovascular

* LVEF normal by echocardiography or radionuclide angiocardiography

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 2 years after study participation
* No psychological, familial, sociological, or geographical condition that would preclude study compliance or follow-up
* No active infection requiring specific therapy (e.g., antibiotics or anti-HIV therapy)
* No other prior or concurrent primary malignant tumor except adequately treated carcinoma in situ of the cervix or squamous cell or basal cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* More than 2 weeks since prior immunotherapy

Chemotherapy

* See Disease Characteristics
* Prior systemic chemotherapy allowed provided all of the following conditions are met:

  * Cumulative anthracycline dose is less than 200 mg/m^2
  * No allergy to anthracyclines
  * Prior methotrexate is low dose (i.e., weekly dose less than 30 mg)
* More than 2 weeks since prior chemotherapy

Endocrine therapy

* See Disease Characteristics
* No concurrent systemic steroids

Radiotherapy

* More than 2 weeks since prior radiotherapy

Surgery

* Not specified

Other

* Recovered from toxic effects of prior therapy, excluding alopecia
* No other concurrent anticancer therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2003-10; Primary Completion 2009-07 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Response (complete clinical [CCR] and partial resp. [PR]) rate by Tumor Burden Index for cutaneous disease and appearance or disappearance of lesions for noncutaneous disease every 8 wks during treatment and then every 12 wks until progression

SECONDARY OUTCOMES:
Time to progression measured by Tumor Burden Index for cutaneous disease and appearance or disappearance of lesions for noncutaneous disease every 8 weeks during treatment
Duration of response measured by Tumor Burden Index for cutaneous disease and appearance or disappearance of lesions for noncutaneous disease every 8 weeks during treatment and then every 12 weeks until progression
Toxicity assessed by CTC v.2.0 at the end of each course

CONTACTS AND LOCATIONS:
Overall Officials: Reinhard Dummer, MD, Study Chair — UniversitaetsSpital Zuerich
Locations (11):
- Austria (2):
  - Karl-Franzens-University Graz, Graz
  - Allgemeines Krankenhaus - Universitatskliniken, Vienna
- Germany (5):
  - Universitaetsklinikum Essen, Essen
  - Klinikum der Friedrich-Schiller Universitaet Jena, Jena
  - Klinikum der Stadt Mannheim, Mannheim
  - Klinikum Minden, Minden
  - Julius Maximilians Universitaet Hospital, Würzburg
- Rambam Medical Center, Haifa, Israel
- Universita di Torino, Turin, Italy
- UniversitaetsSpital Zuerich, Zurich, Switzerland
- St. Thomas' Hospital, London, England, United Kingdom

REFERENCES:
- [Derived] Dummer R, Quaglino P, Becker JC, Hasan B, Karrasch M, Whittaker S, Morris S, Weichenthal M, Stadler R, Bagot M, Cozzio A, Bernengo MG, Knobler R. Prospective international multicenter phase II trial of intravenous pegylated liposomal doxorubicin monochemotherapy in patients with stage IIB, IVA, or IVB advanced mycosis fungoides: final results from EORTC 21012. J Clin Oncol. 2012 Nov 20;30(33):4091-7. doi: 10.1200/JCO.2011.39.8065. Epub 2012 Oct 8. PMID 23045580